CLINICAL TRIAL: NCT04273087
Title: Characterization of a Clinical Subpopulation With Autism Spectrum Disorder
Status: Completed | Type: Observational
Sponsor: Stalicla SA (Industry)
Responsible Party: Sponsor
Other Study IDs: STP1-C003
Record Dates: First submitted 2020-02-06; First posted 2020-02-17 (Actual); Last update posted 2022-11-18 (Actual); Status verified 2022-11

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Observation — Clinical signs and symptoms

SUMMARY:
The main objective for this research study is to gather additional information to help confirm identification of new subgroups within the autism spectrum.

ELIGIBILITY:
Inclusion Criteria:

* Participants previously diagnosed with ASD (DSM-5) supported by either autism diagnostic interview revised (ADI-R) or Autism Diagnostic Observation Scale (ADOS-2) scores
* Available health records within the first 2 years of life
* Participants must have a parent or reliable caregiver who agrees to provide information about the participant

Exclusion Criteria:

* Genetically identified ASD (syndromic form of autism, e.g. fragile X)
* Episode of fever (i.e. ≥100.5 °F) or clinically significant illness without fever (as judged by the Investigator), within 10 days before the study visit

Ages: 10 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Cincinnati Children's Hospital Primary Care Clinic
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Prevalence of non-behavioral phenotypical traits in sub-populations with Autism Spectrum Disorder (ASD) | Day 0
  A questionnaire will be administered to collect non-behavioral traits and co-occurring conditions data of the participants

CONTACTS AND LOCATIONS:
Overall Officials: Craig A Erickson, MD, Principal Investigator — CCHMC
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States